CLINICAL TRIAL: NCT04796142
Title: An Integrated Model to Increase Medication Recognition and Reconciliation in Oncologic Patients
Brief Title: Medication Reconciliation in Oncologic Patients
Acronym: PROF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRST 100.40
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Medication Reconciliation
Keywords: Medication reconciliation; IT platform; Pharmacies
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reconciliation (Experimental): Interventional trial without drugs
  Interventions: Other: medication reconciliation

INTERVENTIONS:
Other: medication reconciliation — medication reconciliation

SUMMARY:
To improve medication reconciliation in oncologic patients in healthcare transitions through an alliance between a Cancer Institute and the community pharmacies and a new integrated IT platform.

DETAILED DESCRIPTION:
This trial will explore the alliance between a Cancer Institute and the community pharmacies to improve medication reconciliation in healthcare transitions, and will validate a new integrated IT platform.

Cancer patients receiving an oncologic treatment will be asked to choose a pharmacy participating to the trial, and to perform the pharmacological survey before every cycle of chemotherapy.

This will be sent through the new IT platform to the electronic medical record of IRST, and the Oncologist will perform the reconciliation.

Data about concomitant medications and possible interactions will be exensively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Patients receiving an anticancer treatment
* Clear understanding of the Italian language; written informed consent.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
medication recognition and reconciliation maintenance | At day 1 of each cycle of treatment (each cycle might be 14, 21 or 28 days)
  number of reconciliations per patient

CONTACTS AND LOCATIONS:
Overall Officials: martina minguzzi, Principal Investigator — IRCCS IRST
Locations (1):
- Alessandro Passardi, Meldola, FC, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Passardi A, Serra P, Donati C, Fiori F, Prati S, Vespignani R, Taglioni G, Farfaneti Ghetti P, Martinelli G, Nanni O, Altini M, Frassineti GL, Minguzzi MV. An Integrated Model to Improve Medication Reconciliation in Oncology: Prospective Interventional Study. J Med Internet Res. 2021 Dec 20;23(12):e31321. doi: 10.2196/31321. PMID 34932001